CLINICAL TRIAL: NCT02923479
Title: Robot-assisted Ankle Rehabilitation Using the High-performance Robotic Device IIT-ARBOT: A Pilot Randomised Controlled Study
Brief Title: Robot-assisted Rehabilitation of Ankle Fractures: Efficacy and Comparison With Traditional Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRMINAIL01
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Ankle Fractures
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: ARBOT Group (Experimental): The patients in the "ARBOT Group" underwent to following interventions:
  1. General Rehabilitation
  2. Specific ankle rehabilitation by ARBOT device
  Interventions: Device: Specific ankle rehabilitation by ARBOT device; Other: General Rehabilitation
- Control Group (Other): The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation
  2. Specific ankle rehabilitation performed by physiotherapist
  3. Specific ankle rehabilitation by Biodex System 3 dynamometer
  4. Specific ankle rehabilitation by ProKin PK254 platform.
  Interventions: Other: General Rehabilitation; Other: Specific ankle rehabilitation performed by physiotherapist; Device: Specific ankle rehabilitation by Biodex System 3 dynamometer; Device: Specific ankle rehabilitation by ProKin PK254 platform

INTERVENTIONS:
Device: Specific ankle rehabilitation by ARBOT device — ARBOT is a programmable robotic device consisting in a two-degree-of-freedom electromechanical platform developed by Italian Institute of Technology - Advanced Robotics and Rehab Technologies. It is composed of a fixed base, a central strut, a moving platform supporting patient's foot and three actuated limbs with a universal-prismatic-spherical kinematic chain. A six-axis force/torque sensor mounted between the moving platform and the footplate senses the human-robot interaction force and torque. The device is interfaced to a standard all-in-one touch screen Personal Computer with graphic applications to give patients visual feedback in real time.
  Arms: Experimental: ARBOT Group
Other: General Rehabilitation — All patients underwent general rehabilitation (gait training, aerobic conditioning), including - if necessary - an initial weight training phase before the functional full weight-bearing program.
Other: Specific ankle rehabilitation performed by physiotherapist — Subjects in the control group underwent manually assisted range of motion exercises.
  Arms: Control Group
Device: Specific ankle rehabilitation by Biodex System 3 dynamometer — Subjects in the control group performed non-robotic resistive training using a Biodex System 3 dynamometer
  Arms: Control Group
Device: Specific ankle rehabilitation by ProKin PK254 platform — Subjects in the control group performed non-robotic proprioceptive training using a ProKin PK254 mobile electronic platform.
  Arms: Control Group

SUMMARY:
The purpose of this trial is to determine the effectiveness, safety and tolerability of robot-assisted rehabilitation using ARBOT in patients with ankle dysfunction resulting from work related ankle fractures, compared with conventional rehabilitation programs.

DETAILED DESCRIPTION:
INTRODUCTION:

Robotic devices for lower-limb rehabilitation have been mainly tested in neurologically injured patients. Up to now, clinical studies using robotic training in orthopedic conditions are few. A pilot study was carried out at INAIL Physical Rehabilitation Center of Volterra using ARBOT, a prototypal robotic system for ankle rehabilitation. This device has been developed by IIT - Italian Institute of Technology and it consists of a two-degree-of-freedom electromechanical platform which is able to perform most of the exercises foreseen by the standard rehabilitation programs. By virtue of its innovative motion system and control architecture, ARBOT integrates multiple rehabilitation equipment functions, performing also special exercise programs such as elastic and fluid-dynamic resistance.

ARBOT allows training according to programmed sequences, in order to promote range of movement, muscular function and proprioceptive recovery. Exercises can be performed with or without bearing weight. Moreover, ARBOT is a powerful evaluation instrument for physiotherapists in order to verify and record the results of rehabilitative intervention.

The primary aim of this trial was to determine the effectiveness, safety and tolerability of robot-assisted rehabilitation using ARBOT in patients with ankle dysfunction resulting from work related ankle fractures, compared with conventional rehabilitation programs. Secondary objectives was to investigate correlations among physical and disability parameters, to collect data in order to define further study protocols and improve ARBOT's performance and ergonomics, and ultimately to evaluate patient satisfaction with respect to robot assisted rehabilitation programs.

METHODS:

Thirty-two patients with work related injuries resulting in ankle and/or hindfoot fractures and subsequent to the immobilization phase was enrolled in an open randomized controlled trial over a 30 month period. Each participant was randomly allocated to experimental or control group and received a 4-week rehabilitation program (20 sessions, for 5 days/week from admission to discharge in the Rehabilitation Centre) and weekly robotic and clinical assessments.

Subjects in the experimental group were treated using ARBOT with passive, active and active assisted range-of-motion exercises, resistive exercises in isometric, isotonic, isokinetic, elastic and fluid-dynamic conditions, and proprioceptive training. Control subjects were assisted by a physiotherapist during range of motion recovery exercises and performed resistive and proprioceptive training using Biodex System 3 dynamometer and ProKin PK254 mobile electronic platform.

The assessment sessions included measurements of dorsiflexion ROM, isometric and isokinetic plantar-flexion torque and proprioceptive performance with ARBOT and 2 minutes walking and timed stair climbing test, LEFS-Lower Extremity Functional Scale and AOFAS-Ankle-Hindfoot Scale.

Site monitoring of the study has been conducted according to the standard ISO 14155.

ELIGIBILITY:
Inclusion Criteria:

1. Functional limitation following work-related ankle injuries, including:

   * Malleolar and/or tibial shaft fractures, both surgically and conservatively treated;
   * Distal tibia and fibula fractures, both surgically and conservatively treated;
   * Hindfoot (Calcaneus and Talus) fractures, both surgically and conservatively treated.
2. Post-immobilization phase;
3. Time interval since fracture event of less than 12 months;
4. Signed informed consent acquisition.

Exclusion Criteria:

1. Non-compliance with study requirements;
2. Pregnancy or breast feeding;
3. Current or prior history of malignancy;
4. Open skin at the level of the patient-device interface;
5. Sensory deficit at the level of the patient-device interface;
6. Ankle motor deficit secondary to peroneal or tibial neuropathy;
7. Acute inflammatory arthritis of the ankle;
8. Other pathological conditions inducing lower limb pain or disfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of Dorsiflexion Range of Motion | At baseline and after 1, 2, 3 and 4 weeks intervention
Change of Isometric peak torque at 0° and 10° of plantar flexion | At baseline and after 2 and 4 weeks intervention
Change of Isokinetic plantar-flexion torque at speed of 30°, 60°, 120°/sec | At baseline and after 2 and 4 weeks intervention
Change of 2 Minute Walk Test (2MWT) | At baseline and after 2 and 4 weeks intervention
Side Effects using ARBOT | Through study completion, up to 4 weeks

SECONDARY OUTCOMES:
Timed Stair Climbing Test (10 steps) | At baseline and after 2 and 4 weeks intervention
Proprioceptive tests (time taking and accuracy) | At baseline and after after 2 and 4 weeks intervention
Pain (VAS 0-10) | At baseline and after 1, 2, 3 and 4 weeks intervention
LEFS - The Lower Extremity Functional Scale | At baseline and after after 4 weeks intervention
AOFAS - Ankle-Hindfoot Scale | At baseline and after 4 weeks intervention
Patient Satisfaction (VAS 0-10) | After 4 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Catitti, MD, Principal Investigator — INAIL - Centro di Riabilitazione Motoria di Volterra
Locations (1):
- INAIL - Centro di Riabilitazione Motoria di Volterra, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saglia JA, Tsagarakis NG, Dai JS, Caldwell DG. Control Strategies for Patient-Assisted Training Using the Ankle Rehabilitation Robot (ARBOT). IEEE ASME TRANSACTIONS ON MECHATRONICS 2013; PP (99): 1-10.
- [Background] Saglia JA, Tsagarakis NG, Dai JS, Caldwell DG. A high-performance redundantly actuated parallel mechanism for ankle rehabilitation. International Journal of Robotics Research 2009; 28 (9): 1216-1227.
- [Background] Saglia JA, Tsagarakis NG, Dai JS, Caldwell DG. Inverse-Kinematics-Based Control of a Redundantly Actuated Platform for Rehabilitation. Journal of Systems and Control Engineering, IMechE Proceedings 2009; 223 (1): 53-70.